CLINICAL TRIAL: NCT00615186
Title: A Phase III Randomized Study of Neuradiab in Combination With External Beam Radiation and Temozolomide Versus External Beam Radiation and Temozolomide in Patients With Newly Diagnosed Glioblastoma Multiforme
Brief Title: Glioblastoma Multiforme (GBM) Locoregional Agent Survival Study - Anti-tenascin Radiolabeled Antibody Therapy
Acronym: Glass-Art
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to delay in site initiation and funding considerations
Sponsor: Bradmer Pharmaceuticals Inc. (Industry)
Responsible Party: David A. Reardon, MD, Duke University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRAD-301
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: Glioblastoma Multiforme
Keywords: Neuradiab; Locoregional glioblastoma multiforme disease; Anti-tenascin; Radiolabeled antibody therapy; Survival
MeSH Terms: conditions — Glioblastoma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Prior Surgery
  Rickham Catheter placement 99mTc-DTPA Flow Study
  Neuradiab Dosimetry Study
  Neuradiab Therapeutic Dose Administration
  Radiation Therapy (XRT) + Temozolomide:
  XRT 5 days/week + temozolomide (75 mg/m2/day) over 6.5 weeks.
  Post-Radiation Temozolomide Therapy:
  Temozolomide 150-200 mg/m2/day × 5 days, every 28 days until patient's death, confirmed disease progression, unacceptable toxicity, non-compliance with the protocol, withdrawal of consent, and/or other factor that in the opinion of the consulting oncologist precludes continued study treatment.
  Interventions: Drug: Neuradiab + Radiotherapy + Temozolomide
- B (Active Comparator): Prior Surgery: Gross total resection (< 1 cm. enhancing rim)
  Radiation Therapy (XRT) + Temozolomide:
  XRT 5 days/week + 42 days of temozolomide (75 mg/m2/day) over 6.5 weeks
  Post-Radiation Temozolomide Therapy:
  Temozolomide 150-200 mg/m2/day × 5 days, every 28 days until patient's death, confirmed disease progression, unacceptable toxicity, non-compliance with the protocol, withdrawal of consent, and/or other factor that in the opinion of the consulting oncologist precludes continued study treatment.
  Interventions: Drug: Radiation Therapy + Temozolomide

INTERVENTIONS:
Drug: Neuradiab + Radiotherapy + Temozolomide — Prior Surgery
  Rickham Catheter placement 99mTc-DTPA Flow Study
  Neuradiab Dosimetry Study
  Neuradiab Therapeutic Dose Administration
  Radiation Therapy (XRT) + Temozolomide:
  XRT 5 days/week + temozolomide (75 mg/m2/day) over 6.5 weeks.
  Post-Radiation Temozolomide Therapy:
  Temozolomide 150-200 mg/m2/day × 5 days, every 28 days until patient's death, confirmed disease progression, unacceptable toxicity, non-compliance with the protocol, withdrawal of consent, and/or other factor that in the opinion of the consulting oncologist precludes continued study treatment.
  Arms: A
Drug: Radiation Therapy + Temozolomide — Prior Surgery: Gross total resection (< 1 cm. enhancing rim)
  Radiation Therapy (XRT) + Temozolomide:
  XRT 5 days/week + 42 days of temozolomide (75 mg/m2/day) over 6.5 weeks
  Post-Radiation Temozolomide Therapy:
  Temozolomide 150-200 mg/m2/day × 5 days, every 28 days until patient's death, confirmed disease progression, unacceptable toxicity, non-compliance with the protocol, withdrawal of consent, and/or other factor that in the opinion of the consulting oncologist precludes continued study treatment.
  Other Names: Temodar (US)
  Arms: B

SUMMARY:
The current study will investigate whether the addition of Neuradiab to surgery, radiation and adjuvant chemotherapy (temozolomide) will improve the survival of patients with glioblastoma and whether the drug regimen is safe.

DETAILED DESCRIPTION:
In all cases where surgery is a possibility, tumor removal is usually indicated as the first step of therapy for glioblastomas. The goals of such surgery include removal of as much tumor mass as possible and preparation of the tumor bed for adjuvant therapy. Except for deaths arising from adverse surgical events (about 1-2% of surgeries), tumor removal enhances survival times. Unfortunately, without additional therapies, most GBM will recur at or near the original tumor site within several months. Addition of radiotherapy to surgery as part of the treatment regimen enhances survival in most patients compared to surgery alone.

The use and benefits of adjuvant chemotherapy for GBM is controversial. Some studies suggest an enhancement of survival from the use of agents such as carmustine (BCNU) and cisplatin, but generally only about 10-20% of the patient population shows such responses (Stewart 2002). The blood-brain barrier presents a major obstacle to traditional uses of chemotherapy in GBM, and, therefore, some clinical trials are focused on delivery of such agents directly to the brain/tumor mass via catheters with pressure-driven infusion.

At present, only two pharmacologic therapies are approved for the treatment of GBM, Gliadel® and Temodar®. Implantation of BCNU-impregnated wafers (Gliadel Wafer, Guilford Pharmaceuticals, approved by the U.S. Food and Drug Administration (FDA) in 1996) after surgery and radiotherapy was the first pharmacologic-chemotherapeutic therapy for GBM. It has shown very modest enhancements in overall survival (11.6 vs. 13.9 months) when added to a regimen of surgery and radiotherapy (Westphal et al. 2006). In this patient population, these agents demonstrate the typical side effects associated with antineoplastic chemotherapies, and are, therefore, often contraindicated. Nevertheless, despite FDA approval and availability of Gliadel for nearly a decade, its utility remains controversial and it is not routinely used in daily clinical practice. In 2005, the FDA approved the use of temozolomide (Temodar ®, Schering-Plough) given concurrently during and subsequent to radiotherapy for the treatment of newly diagnosed GBM. In a multicenter Phase III trial of 573 GBM patients, radiation alone gave a median survival rate of 12.1 months; the addition of temozolomide led to a median survival of 14.6 months (Stupp et al. NEJM 2005). More importantly, the 2-year survival rate increased from 10% with initial radiation alone to 27% with combined chemo- and radiotherapy. This regimen is considered the standard of care for all patients with newly diagnosed glioblastoma. Ongoing clinical trials are exploring alternative temozolomide administration schedules or combination of this regimen with novel chemotherapy or targeted anti-tumor agents assessing the efficacy of temozolomide alone or in various chemotherapeutic combinations are underway (Herrlinger et al. 2006, Mirimanoff et al. 2006, Stupp et al. 2006, Hau et. al. 2007).

The current study will investigate whether the addition of Neuradiab to surgery, radiation and adjuvant chemotherapy (temozolomide) will improve the survival of patients with glioblastoma and whether the drug regimen is safe. Earlier trials have demonstrated that patient-specific dosimetry yields the best combination of safety and efficacy and will be employed in the current trial. The anti-tenascin monoclonal antibody will bind to tenascin glycoprotein associated with residual neuroblastoma cells, causing the associated radioactive iodine to be fixed in close proximity to the tumor delivering cytocidal local radiotherapy. In this way, it is anticipated that residual tumor cells, which represent the primary reason for treatment failure using conventional therapy, will be destroyed, thus prolonging patient survival. The surgery, radiotherapy, and adjuvant chemotherapy will be administered to the patients in the control arm and represents appropriate therapy for this disorder. In addition, tumor samples will be analyzed for methyl guanine methyl transferase (MGMT) activity to see whether the previously observed and reported correlation with outcome is once again observed (Hegi et. al. 2005).

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed supratentorial unifocal lesion seen on magnetic resonance imaging (MRI).
* Patient must have undergone a gross total surgical resection of the tumor mass with post surgical MRI (performed within 14 days of randomization) demonstration of adequacy defined as < 1.0 cm of residual enhancement away from resection cavity perimeter.
* Histopathologically confirmed diagnosis of glioblastoma (World Health Organization [WHO] grade IV astrocytoma) and tumor sample is available. (http://rad.usuhs.mil/rad/who/who2b.html)
* Age ≥ 18 years of age at the time of study entry.
* Karnofsky Performance Status ≥ 60%.
* Adequate bone marrow function, defined as:

  1. Absolute neutrophil count ≥ 1500 cells/mm3
  2. Hemoglobin ≥ 10 g/dL
  3. Platelet count ≥ 100,000 cells/mm3
* Adequate hepatic function, defined as:

  1. Bilirubin ≤ 1.5 mg/dL
  2. SGOT ≤ 2.5 × upper limit of normal (ULN
* Adequate renal function, defined as creatinine ≤ 1.3 mg/dL (µmol/L)
* Patients must have a negative HAMA (human anti-murine antibody) assay.
* Women of childbearing potential must have a negative pregnancy test (serum or urine).
* Men and women of reproductive potential must agree to use an effective contraceptive method including one of the following: surgical sterilization (tubal ligation for women or vasectomy for men); approved hormonal contraceptives (such as birth control pills, Depo-Provera or Lupron Depro); barrier methods (such as condom or diaphragm) used with a spermicide cream or an intrauterine device (IUD).
* Patient must give written informed consent prior to any study-specific procedures being implemented.

Exclusion Criteria:

* Infratentorial tumor, tumor with subependymal spread, multifocal tumor, tumor with ventricular communication, intraventricular tumor or tumor which abuts the motor strip or exceeds beyond the cranial vault.
* Pregnant or lactating females.
* Women of childbearing potential and men who are sexually active and not willing/able to use medically acceptable forms of contraception.
* No severe, active comorbidity, including any of the following:

  1. Unstable angina and/or congestive heart failure requiring hospitalization
  2. Transmural myocardial infarction within the last 6 months
  3. Acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization
  4. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of randomization
  5. Known hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
  6. Known AIDS based upon current CDC definition
  7. Major medical illnesses or psychiatric impairments that, in the investigator's opinion, will prevent administration or completion of protocol therapy
  8. Active connective tissue disorders, such as lupus or scleroderma that, in the opinion of the treating physician, may put the patient at high risk for radiation toxicity.
* Prior or planned chemotherapy, immunotherapy, biologic therapy, radiation therapy, radioimmunotherapy, hormonal therapy, or experimental therapy for brain tumor. Prior or active corticosteroid therapy is permitted.
* History of severe allergic reaction to contrast media.
* Any serious medical condition or psychiatric illness unresponsive to medical intervention.
* Prior malignancy if active treatment was required during the previous 3 years except for adequately treated basal cell or squamous cell skin cancer and in situ uterine cervical cancer.
* Known hypersensitivity to murine proteins.
* Inability to undergo an MRI.
* Patients treated on any other therapeutic clinical trial within 30 days prior to study entry or during participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-06; Primary Completion 2013-08 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
The primary measure of efficacy is overall survival (OS). | Death from any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) is the sole secondary measure of efficacy. | Difference between the date of randomization and the first date of meeting objective criteria for disease progression or death, whichever event is earliest.

CONTACTS AND LOCATIONS:
Overall Officials: David A. Reardon, MD, Principal Investigator — Duke University; Philip J Bierman, MD, Principal Investigator — University of Nebraska; Ray M. Chu, MD, Principal Investigator — Cedars-Sinai Medical Center; Susan C. Pannullo, MD, Principal Investigator — New York Presbyterian - Cornell; Frank D. Vrionis, MD, MPH, PhD, Principal Investigator — Moffitt Cancer Center